CLINICAL TRIAL: NCT00527228
Title: Deflazacort in Dysferlinopathies (LGMD2B/MM) - a Double Blind, Placebo-controlled Clinical Study
Brief Title: Deflazacort in Dysferlinopathies
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Maggie Walter, Prof. Dr. Maggie C. Walter, MD, MA, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 274/02
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: LGMD2B; Miyoshi Myopathy; Dysferlinopathy
Keywords: Muscular dystrophy; therapy; steroids; deflazacort; dysferlinopathy; LGMD; MM
MeSH Terms: conditions — Limb-girdle muscular dystrophy, type 2B; Miyoshi myopathy; Dysferlinopathy; Muscular Dystrophies | interventions — deflazacort; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): After 6 months of treatment, and a 3-months wash-out, there is cross-over to Arm B
  Interventions: Drug: deflazacort
- B (Placebo Comparator): After 6 months of treatment, and a 3-months wash-out, there is cross-over to Arm A
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: deflazacort — In the first 12 months, patients will receive no treatment to assess the natural history of the disease. Afterwards, patients will be treated with deflazacort 1mg/kg/day or placebo for the first month on treatment, from the second month on deflazacort or placebo will be administered on an alternate day regimen). Patients will be randomized to six months verum or placebo each, after a 3-months wash-out patients cross over to the alternate treatment for six months. In a 2-years follow-up phase after the double-blind treatment phase, long-term development of the disorder will be documented.
  Other Names: Calcort; Corticosteroid
  Arms: A
Drug: placebo
  Arms: B

SUMMARY:
The present study is designed to assess the natural history in a one year pre-phase of the trial and evaluate therapeutic efficacy and side effects of deflazacort in LGMD2B/MM patients in a placebo-controlled trial. Furthermore, long-term development of the disease under naturalistic conditions will be documented in a 2-year follow-up after the end of the double-blind treatment phase.

DETAILED DESCRIPTION:
Limb girdle muscular dystrophies (LGMDs) are a genetically heterogeneous group of disorders encompassing various genetically defined subtypes (LGMD 2A-2H). Therapeutic trials should address each disease entity separately to assess effectiveness of medical treatments. A placebo-controlled trial in patients with dysferlinopathy may reveal insights in the natural course of the disease and show therapeutic options in a homogeneous group of patients. So far, steroids are the only drugs showing efficacy in muscular dystrophies, mainly in Duchenne muscular dystrophy (DMD). Both dystrophin and dysferlin are attached to the sarcolemma and deficiency of both proteins cause sarcolemmal defects; therefore, any membrane-stabilizing steroid effect may be beneficial in both DMD and LGMD2B/ Myoshi myopathy (MM). Furthermore, there is marked inflammation in muscle biopsies of many LGMD2B patients. Therefore, the anti-inflammatory effect of steroids may improve muscle function in LGMD2B/MM. In our trial, effects of deflazacort in patients with dysferlinopathy (LGMD2B/MM) on strength and daily-life activities are addressed. The present study is designed to assess the natural history and evaluate therapeutic efficacy and side effects of deflazacort / placebo in LGMD2B/MM patients.

Although no major therapeutic breakthrough has been achieved and curative treatment modalities are not yet applicable, life expectancy and quality of life of dysferlinopathy patients could be remarkably improved by establishing a drug therapy, capable of delaying the dystrophic process and improving muscle strength and function. Therefore, the results of this study are warranted and may influence further guidelines for steroid treatment in dysferlinopathies. Furthermore, the assessment of the natural history of the disease will provide new insights in the clinical understanding of dysferlinopathies.

ELIGIBILITY:
Inclusion Criteria:

* Clinically, histologically, immunohistochemically and genetically defined muscular dystrophy with dysferlin-deficiency (LGMD2B/MM).
* Patients should fulfill clinical, morphological, immunohistochemical and immunoblot criteria of LGMD 2B and definite mutation in dysferlin gene.
* There is no limitation on age for study inclusion.

Exclusion Criteria:

* Patients confined to bed or wheelchair.
* Patients with other neurologic or internistic diseases and patients with former or current steroid treatment will not be included.
* Exclusion criteria during the trial are withdrawal of informed consent or lack of compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-09; Primary Completion 2008-04 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Muscle strength according to Medical Research Council Scales (MRC) and quantitative strength measurement evaluated by hand-held dynamometry (Citec, Groningen, The Netherlands)in the same muscle groups. | each 6 months

SECONDARY OUTCOMES:
Quantitative strength measurement (QSM, M3diagnos, Fa. Schnell, Germany), Neuromuscular Symptoms Score (NSS), timed function tests, Clinical Global Impressions (CGI) of change and quality of life assessment(SF-36 scale). | each 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maggie C. Walter, MD, Principal Investigator — Friedrich-Baur-Institute, Dept. of Neurology, Ludwig-Maximilians-University of Munich, Germany
Locations (1):
- Friedrich-Baur-Institute, Dept. of Neurology, Ludwig-Maximilians-University of Munich, Munich, Germany

REFERENCES:
- [Derived] Walter MC, Reilich P, Thiele S, Schessl J, Schreiber H, Reiners K, Kress W, Muller-Reible C, Vorgerd M, Urban P, Schrank B, Deschauer M, Schlotter-Weigel B, Kohnen R, Lochmuller H. Treatment of dysferlinopathy with deflazacort: a double-blind, placebo-controlled clinical trial. Orphanet J Rare Dis. 2013 Feb 14;8:26. doi: 10.1186/1750-1172-8-26. PMID 23406536
- See also: Homepage of the German Muscular Dystrophy Network (MD-NET) — http://www.md-net.org